CLINICAL TRIAL: NCT03973944
Title: Restoration of Atrioventricular Coupling by Cardiac Resynchronization Therapy in Heart Failure Patients With Prolonged PR Interval
Brief Title: ReachPR Trial Resynchronization Therapy in Heart Failure Patients With Prolonged PR Interval
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL60764.068.17
Record Dates: First submitted 2019-05-31; First posted 2019-06-04 (Actual); Last update posted 2019-08-14 (Actual); Status verified 2019-05

CONDITIONS: Atrioventricular Dyssynchrony; Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Cardiac Resynchronization Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiac resynchronization therapy (Other): AV coupling by atrio-biventricular pacing
  Interventions: Device: Cardiac resynchronization therapy

INTERVENTIONS:
Device: Cardiac resynchronization therapy — Atrio-biventricular pacing to shorten the prolonged PR interval

SUMMARY:
Rationale: Prolongation of the electrocardiographic PR interval (PR interval > 200ms; also known as first-degree atrioventricular block) is frequently encountered in clinical practice and is generally considered as a benign sign. However, there is increasing evidence that a prolonged PR interval results in poor hemodynamic performance with elevated left ventricular (LV) end-diastolic pressures evidenced by diastolic mitral regurgitation. Previous studies have also associated a prolonged PR interval with a substantially increased risk of future atrial fibrillation (AF) and pacemaker-implantation, and increased risk of heart failure (HF) hospitalization and death. These risks stress the importance of proper atrioventricular (AV) coupling. Shortening of the PR interval may be especially important in heart failure patients and can be obtained by atrioventricular pacing. A possible adverse effect of ventricular pacing is that it results in ventricular dyssynchrony which may lead to worsening cardiac function. This effect may be prevented by applying atrio-biventricular pacing. Data from several previous (sub)studies have suggested this.

Objective: The purpose of this study is to investigate the acute hemodynamic effects of restoration of atrioventricular coupling by atrio-biventricular pacing in patients with heart failure and prolonged PR interval.

Study design: This study will be a multi-center, exploratory, prospective interventional, nonrandomized acute hemodynamic study, using patients as their own controls.

Study population: The study will enroll 26 patients with symptomatic heart failure, reduced left ventricular ejection fraction (LVEF) (< 35%) and prolonged PR interval (>230ms), but without seriously prolonged QRS duration (<150ms) or left bundle branch block (LBBB) QRS pattern, who are candidates for an implantable cardioverter defibrillator (ICD) device according to current guidelines.

Main study parameters/endpoints: The main study parameter will be the acute hemodynamic change in left ventricular stroke work (SW) during atrioventricular optimization by atrio-biventricular pacing. Secondary parameters will be the acute hemodynamic changes in left ventricular dP/dt|max and left ventricular stroke volume (SV) by invasive measurements and in left ventricular stroke volume, diastolic mitral regurgitation and left ventricular diastolic filling time by echocardiography during atrioventricular optimization by atrio-biventricular pacing.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: The patients are candidates for an ICD device in whom cardiac resynchronization therapy (CRT) can be considered according to current guidelines. Patients in the present study will receive a CRT-defibrillator (CRT-D). The risk and/or complications of the CRT-D implantation are not additional for this study. After the implantation, acute invasive hemodynamic measurements will be performed with a pressure-volume catheter, which is inserted via the femoral artery and adds approximately 30 minutes to the standard procedure. An extra radiation dose of approximately 50mGy is needed to place the pressure volume catheter in the LV cavity. Local vascular complications of femoral artery puncture like bleeding or damage to the vessel wall may occur but are rare. The non-invasive echocardiographic protocol one to two weeks after implantation will add approximately 45 minutes to the routine outpatient clinic visit. The patients do not have to visit the clinic outside the routine outpatient clinic visits before and after a CRT-D implantation. The patients will have the potential direct benefit from the procedure, by finding the patient's specific optimal (atrioventricular) settings and thereby reducing above described risks of a prolonged PR interval. In case of a worse hemodynamic performance due to the procedure, the CRT-D will be programmed to back up pacing and there is no harm for the patient outside the above subscribed extra measurements.

ELIGIBILITY:
Inclusion Criteria:

* Indication for an ICD device according to current guidelines (24);
* Stable prolonged PR interval >230ms;
* LVEF (< 35%);
* New York Heart Association (NYHA) functional class II, III or ambulant IV;
* Stable sinus rhythm (no documented AF-episodes during the last 4 weeks prior to inclusion);
* Optimal HF (oral) medication, and on a stable medication scheme at least 1 month prior to enrolment; (2)
* Age ≥ 18 years and < 80 years.

Exclusion Criteria:

* Already implanted with an CRT device;
* Resting Heart rate >90 bpm;
* Left bundle branch block (LBBB) QRS morphology;
* QRS duration >150ms
* Recent myocardial infarction (within 40 days prior to enrolment);
* Recent coronary artery bypass graft or valve surgery (within 90 days prior to enrolment);
* Chronic renal failure requiring dialysis;
* Presence of frequent ventricular premature beats (VPB) (>5% on 24h rhythm monitoring or >2 VPB's on ECG at enrolment);
* Moderate to severe aortic valve stenosis (AVA<1,5) or a mechanical aortic valve;
* No femoral arterial access;
* Second or third degree AV block;
* Life expectancy < 1 year;
* Enrolment in one or more ongoing studies that could influence the results of this study.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2018-06-18 (Actual); Primary Completion 2019-12-13 (Estimated); Study Completion 2020-12-13 (Estimated)

PRIMARY OUTCOMES:
Left ventricular stroke work | Acute measurements (during the cardiac resynchronization therapy device-implantation; duration: approximately 1 hours)
  The acute hemodynamic changes in left ventricular stroke work (SW) during atrioventricular optimization by atrio-biventricular pacing.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Vernooy, MD,PhD, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht University Medical Center, Maastricht, Limburg, Netherlands